CLINICAL TRIAL: NCT00651794
Title: Improving Teamwork for Neonatal Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Eric Thomas, Professor - Internal Medicine, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UL1RR024148-01 (NIH)
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Results first posted 2017-10-19 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-09

CONDITIONS: Teamwork During Neonatal Resuscitation
Keywords: Neonatal Resuscitation; Patient Care Team; Medical Errors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (NRP Curriculum with LFT and no team training) (Active Comparator): Standard Neonatal Resuscitation Program (NRP) curriculum with no team training; simulated resuscitation using low-fidelity simulators for low-fidelity training (LFT)
  Interventions: Behavioral: Standard NRP curriculum; Behavioral: Skills practice with low-fidelity mannequin
- NRP with LFT and team training (Experimental): Standard Neonatal Resuscitation Program (NRP) curriculum + team training; simulated resuscitation using low-fidelity simulators for low-fidelity training (LFT)
  Interventions: Behavioral: Teamwork training; Behavioral: Standard NRP curriculum; Behavioral: Skills practice with low-fidelity mannequin
- NRP with HFT and team training (Experimental): Standard Neonatal Resuscitation Program (NRP) curriculum + team training; simulated resuscitations using high-fidelity simulators for high-fidelity training (HFT)
  Interventions: Behavioral: Teamwork training; Behavioral: Standard NRP curriculum; Behavioral: Skills practice with high-fidelity mannequin

INTERVENTIONS:
Behavioral: Teamwork training — Crew Resource Management (CRM) is an aviation training program mandated for all crew members that teaches human factors concepts, communication skills, and teamwork behaviors that can prevent and manage error. Over the last six years the study team has translated these behaviors to neonatal resuscitation and demonstrated that they can be reliably measured. Adding teamwork instruction to the existing NRP, based upon CRM, may be a method to improve communication, teamwork, and the overall quality of neonatal resuscitation.
  Arms: NRP with HFT and team training; NRP with LFT and team training
Behavioral: Standard NRP curriculum — The existing NRP course, taught to most caregivers in the United States who care for newborns, focuses on teaching the technical aspects of neonatal resuscitation with little attention paid to communication and teamwork.
Behavioral: Skills practice with low-fidelity mannequin
  Arms: Control (NRP Curriculum with LFT and no team training); NRP with LFT and team training
Behavioral: Skills practice with high-fidelity mannequin — SimBaby mannequins (Laerdal Medical Corp, Stavanger, Norway) were used in the high-fidelity skills stations. These mannequins have simulated heart tones, breath sounds, pulses, and cries.
  Arms: NRP with HFT and team training

SUMMARY:
The Neonatal Resuscitation Program (NRP) is the curriculum used to teach providers how to care for newborns in the delivery room. Breakdowns in teamwork and communication contribute to NRP quality problems. Adding teamwork instruction to NRP may be a method to improve communication, teamwork, and the overall quality of neonatal resuscitation. This study uses simulation to incorporate team training into NRP and to evaluate both the effectiveness and duration of the team training. Furthermore, because high fidelity simulation is very expensive and not widely available, we will compare NRP with low fidelity team training to NRP with high fidelity team training.

Our hypotheses are:

1. NRP with low fidelity team training results in a) better teamwork, and b) better quality of care compared with standard NRP.
2. NRP with high fidelity team training does not result in better teamwork or better quality of care than NRP with low fidelity simulation.
3. NRP with high fidelity team training does not produce a longer lasting effect on teamwork than NRP with low fidelity simulation.

ELIGIBILITY:
Inclusion Criteria:

* New interns that enter pediatrics, family medicine, obstetrics/gynecology, and emergency medicine.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-06; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Thomas, MD, MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center, Houston, Houston, Texas, United States

REFERENCES:
- [Background] Thomas EJ, Sexton JB, Helmreich RL. Translating teamwork behaviours from aviation to healthcare: development of behavioural markers for neonatal resuscitation. Qual Saf Health Care. 2004 Oct;13 Suppl 1(Suppl 1):i57-64. doi: 10.1136/qhc.13.suppl_1.i57. PMID 15465957
- [Background] Thomas EJ, Sexton JB, Lasky RE, Helmreich RL, Crandell DS, Tyson J. Teamwork and quality during neonatal care in the delivery room. J Perinatol. 2006 Mar;26(3):163-9. doi: 10.1038/sj.jp.7211451. PMID 16493432
- [Background] Thomas EJ, Taggart B, Crandell S, Lasky RE, Williams AL, Love LJ, Sexton JB, Tyson JE, Helmreich RL. Teaching teamwork during the Neonatal Resuscitation Program: a randomized trial. J Perinatol. 2007 Jul;27(7):409-14. doi: 10.1038/sj.jp.7211771. Epub 2007 Jun 7. PMID 17538634
- [Result] Thomas EJ, Williams AL, Reichman EF, Lasky RE, Crandell S, Taggart WR. Team training in the neonatal resuscitation program for interns: teamwork and quality of resuscitations. Pediatrics. 2010 Mar;125(3):539-46. doi: 10.1542/peds.2009-1635. Epub 2010 Feb 15. PMID 20156896

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All incoming interns for pediatrics, combined pediatrics and internal medicine, family medicine, emergency medicine, and obstetrics and gynecology who began training in June 2007 or June 2008 and had not previously completed NRP certification were eligible for participation in the study.
Pre-assignment Details: 100 interns were consented, and 98 completed the initial megacode (that is, the initial simulation with a mannequin that was observed and scored). Baseline characteristics are reported for the 98 who completed the initial megacode.
Groups:
- Control (NRP Curriculum With LFT and no Team Training): Standard NRP curriculum with no team training; simulated resuscitation using low-fidelity simulators
- NRP With LFT and Team Training: Standard NRP curriculum + team training; simulated resuscitation using low-fidelity simulators
- NRP With HFT and Team Training: Standard NRP curriculum + team training; simulated resuscitations using high-fidelity simulators
Period: Overall Study
Arm/Group | Control (NRP Curriculum With LFT and no Team Training) | NRP With LFT and Team Training | NRP With HFT and Team Training
Started | 36 | 31 | 31
Completed | 15 | 9 | 10
Not Completed | 21 | 22 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (NRP Curriculum With LFT and no Team Training) | NRP With LFT and Team Training | NRP With HFT and Team Training | Total
Number analyzed (Participants) | 36 | 31 | 31 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 36 | 31 | 31 | 98
  >=65 years | 0 | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants]
  Unknown | 36 | 31 | 31 | 98
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 31 | 93

OUTCOME MEASURES:

1. Primary Outcome: Teamwork Event Rate
Description: The teamwork event rate was calculated by summing the number of scored teamwork events (sharing information, inquiry, assertion, teaching/advising, and evaluation of plans) and dividing by the total resuscitation time (in minutes).
Time Frame: During the megacode, which was performed about 1 hour after the training
Measure: Mean (Standard Deviation); unit: teamwork events per minute
Arm/Group | Control (NRP Curriculum With LFT and no Team Training) | NRP With LFT and Team Training | NRP With HFT and Team Training
Number analyzed (Participants) | 36 | 31 | 31
teamwork events per minute | 9 (2.10) | 10.3 (3.30) | 12.8 (3.40)

2. Secondary Outcome: Percentage of Time Spent on Workload Management
Description: Workload management percentage was calculated by summing the total time the team demonstrated workload management behavior and dividing by the total resuscitation time.
Time Frame: During the megacode, which was performed about 1 hour after the training
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Control (NRP Curriculum With LFT and no Team Training) | NRP With LFT and Team Training | NRP With HFT and Team Training
Number analyzed (Participants) | 36 | 31 | 31
percentage of time | 89.4 (15) | 98.0 (5.7) | 98.8 (5.4)

3. Secondary Outcome: Percentage of Time Spent on Vigilance
Description: Vigilance percentage was calculated by summing the total time the team demonstrated vigilance behavior and dividing by the total resuscitation time.
Time Frame: During the megacode, which was performed about 1 hour after the training
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Control (NRP Curriculum With LFT and no Team Training) | NRP With LFT and Team Training | NRP With HFT and Team Training
Number analyzed (Participants) | 36 | 31 | 31
percentage of time | 99.6 (0.8) | 99.7 (1.0) | 99.9 (0.3)

4. Secondary Outcome: Neonatal Resuscitation Program (NRP) Quality as Assessed by NRP Performance Score
Description: We analyzed 2 measures of NRP quality: performance score and resuscitation duration. The performance score was calculated by averaging the scores (ranging from 0 to 2 - higher values represent a better outcome) for each NRP step (some of which occurred multiple times). Those scores were summed and divided by the total possible score (2 times the number of steps that should have been performed). When a step was not indicated for the specific resuscitation scenario (e.g., meconium aspiration), that step was not scored by the observers and it was not included in the denominator for performance calculation. This produced a measure of performance percentage ranging from 0 percent to 100 percent (higher values represent a better outcome) for each resuscitation.
Time Frame: During the megacode, which was performed about 1 hour after the training
Measure: Mean (Standard Deviation); unit: performance percentage
Arm/Group | Control (NRP Curriculum With LFT and no Team Training) | NRP With LFT and Team Training | NRP With HFT and Team Training
Number analyzed (Participants) | 36 | 31 | 31
performance percentage | 71.5 (8.3) | 73.4 (7.6) | 72.4 (9.1)

5. Secondary Outcome: Neonatal Resuscitation Program (NRP) Quality as Assessed by Resuscitation Duration
Description: Resuscitation duration is time required to complete the resuscitation. The total duration for each resuscitation was calculated from the start of the instructor's reading of the scenario to the team's statement that the infant should be transferred to the NICU. When any teaching moments occurred during the simulation, the total teaching time was subtracted from the resuscitation duration.
Time Frame: During the megacode, which was performed about 1 hour after the training
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Control (NRP Curriculum With LFT and no Team Training) | NRP With LFT and Team Training | NRP With HFT and Team Training
Number analyzed (Participants) | 36 | 31 | 31
seconds | 634 (259) | 514 (139) | 443 (142)

ADVERSE EVENTS:
Arm/Group | Control (NRP Curriculum With LFT and no Team Training) | NRP With LFT and Team Training | NRP With HFT and Team Training
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/36 | 0/31 | 0/31

LIMITATIONS AND CAVEATS:
Questions remain about whether similar training will be effective for other types of caregivers. Generalizability might be limited if other sites were not able to re-create the team training content.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes